CLINICAL TRIAL: NCT04073472
Title: A Phase I Study of Allogeneic Bone Marrow Derived Mesenchymal Stem Cells for the Treatment of Ileal Anal Anastomosis and Ileal Pouch Fistulas in the Setting of Crohn's Disease of the Pouch
Brief Title: Mesenchymal Stem Cells for the Treatment of Pouch Fistulas in Crohn's
Acronym: IPAAF
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This clinical trial was entered in error. Please refer to the correct entry of this study using the following link: https://clinicaltrials.gov/ct2/show/NCT04519684
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Amy Lightner, Staff Surgeon, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Record Dates: First submitted 2019-08-23; First posted 2019-08-29 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Crohn's Disease; Fistula; Anal Fistula; Pouch, Ileal; Pouches, Ileoanal
Keywords: crohn disease; mesenchymal stem cells; pouch fistulas
MeSH Terms: conditions — Crohn Disease; Fistula; Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mesenchymal stem cells (MSCs) (Experimental): Direct injection of 75 million allogeneic bone marrow derived mesenchymal stem cells (MSC) into ileal pouch fistula at baseline and possibly again after 3 months if not completely healed.
  Interventions: Drug: mesenchymal stem cells (MSCs)

INTERVENTIONS:
Drug: mesenchymal stem cells (MSCs) — Allogeneic bone marrow derived mesenchymal stem cells (MSCs) direct injection to an ileal pouch fistula in the setting of Crohn's disease of the pouch
  Other Names: Allogeneic Bone Marrow Derived Mesenchymal Stem Cells

SUMMARY:
The purpose of this study is to determine the safety and feasibility of using allogeneic bone marrow derived mesenchymal stem cells (MSCs) to treat people with an ileal pouch anal anastomosis (IPAA) who develop a fistula in the setting of Crohn's disease of the pouch.

DETAILED DESCRIPTION:
Proctocolectomy with ileal pouch anal anastomosis (IPAA) remains the procedure of choice for patients with ulcerative colitis (UC). IPAA allows at risk tissue to be removed with restoration of intestinal continuity while maintaining favorable long-term functional outcomes and quality of life. While less than 30% of patients experience short-term postoperative morbidity following IPAA, up to 15% of pouches will ultimately fail due to technical or inflammatory complications, the majority of which manifest as a fistula from the pouch to the perianal or vaginal locations. Pouch failure due to a fistula tract is notoriously difficult to treat. Despite immunosuppressive medications and attempts at local repair, most patients will end up with a pouch excision and permanent ostomy. This can be a devastating outcome in some patients as it impacts body image and quality of life.

Pelvic sepsis following original IPAA has been reported in 5% to 25% of patients, and is the leading cause of pouch failure due to the development of pelvic fibrosis and decreased distensibility of the pouch, ultimately resulting in poor pouch function. One of the leading causes of pelvic sepsis and development of a pouch fistula is Crohn's Disease (CD) of the pouch. While the majority of pouches are constructed for UC, up to 25% of patients with an IPAA will end up having a change in diagnosis from UC to CD or development of de novo CD of the pouch.

The first report of successful healing of a Crohn's fistula with mesenchymal stem cells (MSCs) was in 2003. Since them great enthusiasm has spurred several phase I phase II, and phase III trials designed to study the safety and efficacy of MSCs for perianal CD, all of which have reported encouraging results with regard to safety and efficacy. With over 300 patients now treated, there is a large body of evidence supporting the local delivery of MSCs to heal perianal Crohn's fistulas. Peri-pouch fistulas are similar to Crohn's perianal fistulas except that instead of the rectum containing the internal opening of the fistula, the internal opening is in the ileal pouch, constructed in place of the rectum.

Given the high safety profile and relative success in treating perianal Crohn's disease with mesenchymal stem cells, the investigators are using a GMP grade allogeneic bone marrow derived MSC cell line to establish safety and secondarily monitor for healing in patients with ileal pouch fistulas in the setting of Crohn's disease of the pouch. This trial will use allogeneic bone marrow derived mesenchymal stem cells (MSCs) to produce regenerative signals. The specific rationale for MSCs in IPAA is based upon 1) their anti-inflammatory properties; 2) published experience of MSC in this condition and perianal Crohn's fistula demonstrating efficacy and safety; 3) existence of cGMP methods for their isolation and growth.

This study will enroll adult men and women who have undergone IPAA at least six months prior and now have a peri-pouch fistula related to Crohn's disease of the pouch. Patients who are refractory to conventional medical therapy will be considered. Patients enrolled will be those that meet current indications.

ELIGIBILITY:
Inclusion Criteria

1. Men and women 18-75 years of age who have undergone an ileal pouch anal anastomosis at least 6 months prior who have developed a clinical diagnosis of Crohn's disease of the pouch as determined by a combination of clinical symptoms, pouchoscopy with biopsy, enterography.
2. Single and multi-tract (up to 2 internal and 3 external openings) fistula tract arising from the ileal pouch, ileal anal anastomosis, or anal canal distal to anastomosis that travels to the perianal skin, perineal body, or vagina. Patients with fistulas that arise from the pouch, anastomosis, or anal canal distal to the anastomosis will both be included in enrollment.

   1. Acceptable internal openings and tract locations for the fistula to arise from include the ileal pouch body, the pouch anal anastomosis, and the anal canal distal to the anastomosis.
   2. Acceptable external openings and tract locations for the fistula to arise from include the perianal skin, perineal body, and/or the vaginal wall.
3. Concurrent Crohn's related therapies with stable doses (>3 months) corticosteroids, 5-ASA drugs, immunomodulators, anti-TNF therapy, anti-integrin and anti-interleukin are permitted.
4. Have failed conventional medical therapies described above, defined as a lack of response to systemic immune suppression (e.g. azathioprine, methotrexate, 6-mercaptopurine) or biologic (e.g. anti-TNF, anti-integrin, anti-interleukin) therapies to treat fistulizing CD for at least 3 months
5. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
6. Competent and able to provide written informed consent
7. Ability to comply with protocol.

Exclusion Criteria

1. Inability to give informed consent.
2. Severe antibiotic refractory pouchitis
3. Severe cuffitis refractory to antibiotics
4. Change in medical management for CD in the previous 2 months or changes anticipated in the next 2 months
5. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
6. Specific exclusions;

   1. HIV
   2. Hepatitis B or C
   3. Abnormal CBC at screening
   4. Abnormal AST or ALT at screening
7. History of cancer including melanoma (with the exception of localized skin cancers)
8. Investigational drug within thirty (30) days of baseline
9. Pregnant or breast feeding or trying to become pregnant
10. Branching fistula tract that has > 2 internal openings or 3 external openings,

    1. Patients with greater than 3 blind/branching tracts are excluded
    2. Fistula tracts on the left and/or right side are allowed
11. Allergic to local anesthetics
12. Unwilling to agree to use acceptable contraception methods during participation in study
13. Patients with a non-abscessed chronic cavity will not be included in enrollment
14. Known allergy to DMSO solution

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Feasibility: Number Of Adverse Events | Baseline, Drug administration Visit, Day 1, 1 week, 2 weeks, 1 month, 2 months, 3 month, 6 month, 12 month after each MSCs injection
  Evaluate the number of adverse event occurring during the trial (including clinically significant changes in physical examination, radiographic images, safety lab tests, vital signs).

SECONDARY OUTCOMES:
Radiographic Healing | Baseline, 1 week, 2 weeks, 1 month, 2 months, 3 month, 6 month, 12 month after each 100% cessation of drainage on both clinical exam with deep palpation and per patient MSCs injection
  Number of Participants with:
  Complete Healing MRI with an absence of a fluid collection >2 cm in 3 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Partial Healing MRI with an absence of a fluid collection >2 cm in 2 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Partial Response MRI with an absence of a fluid collection >2 cm in 2 of 3 dimensions, lack of worsening inflammation or new tracts formed
  Lack of Response Radiographic healing which does not meet the threshold for Partial Response
  Decreased symptoms Greater than 50% reduction in drainage as reported by the patient at study visits.
Clinical Healing | Baseline, 1 week, 2 weeks, 1 month, 2 months, 3 month, 6 month, 12 month after each 100% cessation of drainage on both clinical exam with deep palpation and per patient MSCs injection
  Number of Participants with:
  Complete Healing 100% cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
  Partial Healing Greater than or equal to 50 % cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
  Partial Response Less than 50% cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
  Lack of Response Clinical healing which does not meet the threshold for Partial Response
  Decreased symptoms Greater than 50% reduction in drainage as reported by the patient at study visits.

OTHER OUTCOMES:
Alloimmune response to mesenchymal stem cells | Baseline, 1 week, 3 months 12 months after each MSCs injection
  Measure HLA Class I & II SAB Antibody Screening - measures the presence (positive) or absence (negative) of antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lightner, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Background] Cho YB, Lee WY, Park KJ, Kim M, Yoo HW, Yu CS. Autologous adipose tissue-derived stem cells for the treatment of Crohn's fistula: a phase I clinical study. Cell Transplant. 2013;22(2):279-85. doi: 10.3727/096368912X656045. Epub 2012 Sep 21. PMID 23006344
- [Background] Dietz AB, Dozois EJ, Fletcher JG, Butler GW, Radel D, Lightner AL, Dave M, Friton J, Nair A, Camilleri ET, Dudakovic A, van Wijnen AJ, Faubion WA. Autologous Mesenchymal Stem Cells, Applied in a Bioabsorbable Matrix, for Treatment of Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2017 Jul;153(1):59-62.e2. doi: 10.1053/j.gastro.2017.04.001. Epub 2017 Apr 9. PMID 28400193
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Background] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960
- [Background] Molendijk I, Bonsing BA, Roelofs H, Peeters KC, Wasser MN, Dijkstra G, van der Woude CJ, Duijvestein M, Veenendaal RA, Zwaginga JJ, Verspaget HW, Fibbe WE, van der Meulen-de Jong AE, Hommes DW. Allogeneic Bone Marrow-Derived Mesenchymal Stromal Cells Promote Healing of Refractory Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2015 Oct;149(4):918-27.e6. doi: 10.1053/j.gastro.2015.06.014. Epub 2015 Jun 25. PMID 26116801
- [Background] Cho YB, Park KJ, Yoon SN, Song KH, Kim DS, Jung SH, Kim M, Jeong HY, Yu CS. Long-term results of adipose-derived stem cell therapy for the treatment of Crohn's fistula. Stem Cells Transl Med. 2015 May;4(5):532-7. doi: 10.5966/sctm.2014-0199. Epub 2015 Mar 31. PMID 25829404
- [Background] Lee WY, Park KJ, Cho YB, Yoon SN, Song KH, Kim DS, Jung SH, Kim M, Yoo HW, Kim I, Ha H, Yu CS. Autologous adipose tissue-derived stem cells treatment demonstrated favorable and sustainable therapeutic effect for Crohn's fistula. Stem Cells. 2013 Nov;31(11):2575-81. doi: 10.1002/stem.1357. PMID 23404825
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Expanded allogeneic adipose-derived mesenchymal stem cells (Cx601) for complex perianal fistulas in Crohn's disease: a phase 3 randomised, double-blind controlled trial. Lancet. 2016 Sep 24;388(10051):1281-90. doi: 10.1016/S0140-6736(16)31203-X. Epub 2016 Jul 29. PMID 27477896
- [Background] Ciccocioppo R, Bernardo ME, Sgarella A, Maccario R, Avanzini MA, Ubezio C, Minelli A, Alvisi C, Vanoli A, Calliada F, Dionigi P, Perotti C, Locatelli F, Corazza GR. Autologous bone marrow-derived mesenchymal stromal cells in the treatment of fistulising Crohn's disease. Gut. 2011 Jun;60(6):788-98. doi: 10.1136/gut.2010.214841. Epub 2011 Jan 21. PMID 21257987
- [Background] de la Portilla F, Alba F, Garcia-Olmo D, Herrerias JM, Gonzalez FX, Galindo A. Expanded allogeneic adipose-derived stem cells (eASCs) for the treatment of complex perianal fistula in Crohn's disease: results from a multicenter phase I/IIa clinical trial. Int J Colorectal Dis. 2013 Mar;28(3):313-23. doi: 10.1007/s00384-012-1581-9. Epub 2012 Sep 29. PMID 23053677